CLINICAL TRIAL: NCT07226895
Title: A Study to Explore Changes in Cognitive, Clinical, Biological and Digital Measures Following 8 Weeks of Twice-daily Dosing of MT1988 and to Evaluate Safety & Tolerability of MT1988, in Participants at Clinical High Risk (CHR) for Psychosis
Brief Title: A Study Exploring Changes in a Variety of Biomarkers Following Dosing With MT1988 in Participants at Clinical High Risk for Psychosis
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Monument Therapeutics Limited (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Foundation for the National Institutes of Health (Other); ProCAN (Unknown); CT-DPACC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AMP SCZ MT1988 / SCZ201; U01MH137298 (NIH); U24MH137171 (NIH)
Record Dates: First submitted 2025-10-24; First posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Clinical High Risk for Psychosis (CHR)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MT1988 Low Dose (Experimental)
  Interventions: Drug: MT1988 Low Dose
- MT1988 High Dose (Experimental)
  Interventions: Drug: MT1988 High Dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT1988 Low Dose — Oral dosing MT1988; dose level 1
  Arms: MT1988 Low Dose
Drug: MT1988 High Dose — Oral dosing MT1988; dose level 2
  Arms: MT1988 High Dose
Drug: Placebo — Oral Placebo; blinded to match MT1988 all doses
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn how tests undertaken by people at high risk of developing psychosis (aged 17 to 30 years old) change when those people are given the study drug MT1988 daily for 8 weeks. This will help identify tests that could be used in later trials developing treatments for symptoms in people at high risk of developing psychosis, to measure whether those new treatments are effective.

The main question this trial aims to answer is:

Can any of the tests (biomarkers) used in this study detect changes in participants dosed with one of two different dose levels of MT1988?

Researchers will compare the results from two dose levels of MT1988 to a placebo group. Researchers do not expect to see the test results change in participants taking placebo and this will be compared to changes expected in test results in participants taking MT1988.

Participants will:

* take a dose of MT1988 or placebo twice per day for 8 weeks
* attend clinic appointments every two weeks to undertake assessments
* report any side effects they experience to the researchers

ELIGIBILITY:
Inclusion Criteria:

* Aged 17 to 30 years at time of consent.
* Capacity to provide informed consent. (For patients under 17 years, participants must assent and informed consent provided by one parent or legal guardian).
* Meet diagnostic criteria for Clinical High Risk of Psychosis (CHR).
* For females of reproductive potential - not pregnant or nursing and willing to comply with contraceptive requirements.

Exclusion Criteria:

* Clinically significant medical disorder or laboratory test abnormality at Day 1.
* History of or current condition which may prevent participant from complying with study procedures.
* Past or current schizophrenia, other disorder with symptoms of psychosis, major cognitive disorder resulting from traumatic brain injury.
* Received antipsychotic medication equivalent to a total lifetime haloperidol dose >50 mg.
* Current use of medications which could interfere with the study endpoints - to be assessed by the Investigator at screening.
* Unable to abstain from nicotine (e.g. cigarettes, vape) for two hours before cognitive testing.
* Unable to abstain from marijuana use on test day prior to test completion.
* History of suicide attempt or behavior in previous 12 months, or risk of suicidal behavior during the study.

Ages: 17 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to week 8 in test of verbal memory (List Learning Task) as measured by the Penn Computerized Neurobehavioral Battery (PennCNB) test battery | Day 56
Change from baseline to week 8 in attenuated positive symptoms as measured by PSYCHS-CT total score | Day 56
  PSYCHS-CT: Positive Symptoms and Diagnostic Criteria for the Comprehensive Assessment of At-Risk Mental States (CAARMS) Harmonized with the Structured Interview for Pyschosis-risk Syndromes (SIPS) - Clinical Trials version.
  Total score of 0-90 across maximum 15 domain; where a higher score indicates more severe symptoms
Change from baseline to week 8 in negative symptoms as measured by the Negative Symptom Inventory - Psychosis Risk (NSI-PR) total score | Day 56
  Total score of 0-44 across 11 domains; where a higher score indicates more severe symptoms

SECONDARY OUTCOMES:
Safety & tolerability as measured by number of treatment related adverse events | Day 1 to Day 84
  The total number of treatment related adverse events reported per study arm (high dose MT1988, low dose MT1988, placebo) will be compared
Safety & tolerability as measured by proportion of participants with treatment related adverse events | Day 1 to Day 84
  The proportion of participants in each study arm (high dose MT1988, low dose MT1988, placebo) experiencing treatment related adverse events will be compared
Change from baseline to week 4 in test of verbal memory (List learning task) as measured by PennCNB battery | Day 28
Change from baseline to weeks 4 and 8 in overall composite score of cognitive performance as measured by PennCNB test battery | Day 28 and Day 56
  Composite includes Continuous Performance Test, Fractal N-Back, Digit-Symbol Substitution Test, Digit Symbol Recall, Visual Object Learning Test, Emotion Recognition Test, Finger Tapping Test, Motor Praxis
Change from baseline to weeks 4 and 8 in a cognitive test of working memory and executive function as measured by CANTAB SWM test. | Day 28 and Day 56
Change from baseline to weeks 4 and 8 in a cognitive test of sustained attention as measured by CANTAB RVP test. | Day 28 and Day 56
Change from baseline to weeks 4 and 8 in neurophysiology (EEG) as measured by mismatch negativity; auditory oddball P300. | Day 28 and Day 56
Change from baseline to week 4 in attenuated positive symptoms, as measured by the PSYCHS-CT total score. | Day 28
  PSYCHS-CT: Positive Symptoms and Diagnostic Criteria for the Comprehensive Assessment of At-Risk Mental States (CAARMS) Harmonized with the Structured Interview for Pyschosis-risk Syndromes (SIPS) - Clinical Trials version.
  Total score of 0-90 across maximum 15 domain; where a higher score indicates more severe symptoms
Change from baseline to week 4 in negative symptoms as measured by the NSI-PR total score. | Day 28
  Total score of 0-44 across 11 domains; where a higher score indicates more severe symptoms
Change from baseline to weeks 4 and 8 in overall psychopathology as measured by the Positive And Negative Symptoms Scale (PANSS) total score. | Day 28 and Day 56
  Total PANSS score between 30 and 120; where a higher score indicates more severe symptoms
Change from baseline to weeks 4 and 8 in symptoms of anxiety as measured by the Overall Anxiety Severity and Impairment Scale (OASIS). | Day 28 and Day 56
  The OASIS (Overall Anxiety Severity and Impairment Scale) ranges from 0 to 20. Higher scores indicate greater severity and impairment due to anxiety symptoms.
Change from baseline to weeks 4 and 8 in symptoms of depression as measured by the Calgary Depression Scale for Schizophrenia (CDSS). | Day 28 and Day 56
  The Calgary Depression Scale for Schizophrenia (CDSS) ranges from 0 to 27. Higher scores indicate more severe depressive symptoms in individuals with schizophrenia.
Change from baseline to weeks 4 and 8 in symptoms of stress as measured by the Perceived Stress Scale (PSS). | Day 28 and Day 56
  The Perceived Stress Scale (PSS) ranges from 0 to 40. Higher scores indicate greater levels of perceived stress
Change from baseline to weeks 4 and 8 in sleep disturbance as measured by the Patient-Reported Outcomes Measurement Information System - Sleep Disturbance (PROMIS-SD). | Day 28 and Day 56
  The PROMIS-SD scale ranges from 8 to 40. Higher scores indicate greater severity of recent sleep disturbance.
Change from baseline to week 8 in biospecimen assays (levels of inflammation) as measured by blood samples (ELISA). | Day 56
Change from baseline to week 8 in cortisol levels, indicative of stress response, as measured by saliva collection (ELISA). | Day 56
Change from baseline to week 8 in physical/sedentary behavior as measured by a phone accelerometer and assessed by the mindLAMP app | Day -7 to Day 56
Change from baseline to week 8 in roaming/movement behavior as measured by a phone GPS and assessed by the mindLAMP app | Day -7 to Day 56
Change from baseline to week 8 in screen state (screen on/off timestamps) assessed by the mindLAMP app | Day -7 to Day 56
Correlation between latent inhibition score and cognitive change from baseline to weeks 4 and 8 as measured by CANTAB SWM. | Day 28 and Day 56
  The data will be explored to determine whether the score on the latent inhibition assessment tool ("positive", "negative") correlates with cognitive change from baseline to weeks 4 and 8 as measured by CANTAB SWM, using Pearson's correlation coefficient.
Correlation between latent inhibition score and cognitive change from baseline to weeks 4 and 8 as measured by CANTAB RVP. | Day 28 and Day 56
  The data will be explored to determine whether the score on the latent inhibition assessment tool ("positive", "negative") correlates with cognitive change from baseline to weeks 4 and 8 as measured by CANTAB RVP, using Pearson's correlation coefficient.
Correlation between the polygenic risk score (as measured by plasma isolated-DNA samples) and PennCNB score change at week 8. | Day 56
  Polygenic risk scores serve to modestly improve psychosis risk prediction. The data will be examined for correlation between individual genetic risk prediction for psychosis and any changes between baseline and Day 56 for each individual biomarker, using Pearson's correlation coefficient.
Correlation between the polygenic risk score (as measured by plasma isolated-DNA samples) and PYSCHS-CT score change at week 8. | Day 56
  Polygenic risk scores serve to modestly improve psychosis risk prediction. The data will be examined for correlation between individual genetic risk prediction for psychosis and any changes between baseline and Day 56 for each individual biomarker, using Pearson's correlation coefficient.
Correlation between the polygenic risk score (as measured by plasma isolated-DNA samples) and NSI-PR score change at week 8. | Day 56
  Polygenic risk scores serve to modestly improve psychosis risk prediction. The data will be examined for correlation between individual genetic risk prediction for psychosis and any changes between baseline and Day 56 for each individual biomarker, using Pearson's correlation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Woods, M.D., Principal Investigator — Yale University of Medicine; Martha E Shenton, PhD, Principal Investigator — Massachusetts General Brigham
Locations (15):
- United States (15):
  - University of California, Irvine, Irvine, California
  - University of California, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Yale University Conneticut Mental Health Center, New Haven, Connecticut
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Northwell Health, Glen Oaks, New York
  - Columbia University, New York, New York
  - Icahan School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Ohio State University, Columbus, Ohio
  - Prevention Science Institute, Eugene, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
All clinical and phenotypic data will be shared with the NIMH National Data Archive (NDA). All data will be de-identified prior to receipt by the NDA, but the information needed to generate a global unique identifier for the NDA will be collected for each participant. Phenotypic and clinical data will be collected and deposited in the NDA using the data dictionaries available in NDA. Audio files will be transcribed using HIPAA-compliant services. Only pseudo-anonymized transcripts will be sent to the NDA.